CLINICAL TRIAL: NCT06354725
Title: Effect of Weekly Plyometric Training Frequency on Youth Female Basketball Players: A Comparison of Two vs. Four Sessions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bruno Figueira (Other)
Collaborators: Vytautas Magnus University (Other)
Responsible Party: Sponsor-Investigator, Bruno Figueira, Dr., University of Évora
Organization: University of Évora (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2vs4
Record Dates: First submitted 2024-03-21; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Physical Performance
Keywords: physical performance; strength and conditioning; jumps; in-season
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2PLYO (Experimental): The 2PLYO (two-times-a-week) group performed 240 jumps over two sessions (120 jumps per session).
  Interventions: Other: Plyometric
- 4PLYO (Experimental): The 4PLYO (four-times-a-week) group performed 240 jumps over four sessions (60 jumps per session)
  Interventions: Other: Plyometric

INTERVENTIONS:
Other: Plyometric — Players were randomly assigned to a two-times-a-week (2PLYO, n = 15) or four-times-a-week (4PLYO, n = 15) PT group. Both groups performed the same weekly total volume of jumps during PT in addition to regular basketball training and competition. After the eight-week intervention, all players underwent a one-week detraining period with no PT training while basketball training and competitions continued. Testing was performed at baseline (pre-test), after intervention (post-test), and after the detraining period. Players were assessed for lower body power using jump tests (countermovement jump [CMJ], drop-jump [DJ] from a 20-cm box, and horizontal jump [HJ]; change of direction ability using a planned agility test; and speed using a 20-m sprint and a 5-m split.

SUMMARY:
Players were randomly assigned to a two-times-a-week (2PLYO, n = 15) or four-times-a-week (4PLYO, n = 15) PT (Plyometric Training) group. Both groups performed the same weekly total volume of jumps during PT in addition to regular basketball training and competition. The 2PLYO group performed 240 jumps over two sessions (120 jumps per session), and the 4PLYO group performed 240 jumps over four sessions (60 jumps per session). After the eight-week intervention, all players underwent a one-week detraining period with no PT training while basketball training and competitions continued. Testing was performed at baseline (pre-test), after intervention (post-test), and after the detraining period. Players were assessed for lower body power using jump tests (countermovement jump [CMJ], drop-jump [DJ] from a 20-cm box, and horizontal jump [HJ]; change of direction ability using a planned agility test; and speed using a 20-m sprint and a 5-m split.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of four basketball training sessions with at least 90-min duration and one competitive game per week.

Exclusion Criteria:

* Musculoskeletal, neurological, or orthopedic injury that may impair their participation.

Ages: 14 Years to 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Horizontal jump | 10 weeks
  Players performed two jumps for each protocol, with one minute of rest provided between trials and three minutes of rest between protocols. The best result was recorded for analysis.
  In the HJ, a metric tape was used to measure the length between the players' starting position and the nearest point of landing contact (i.e., the back of the heels). The players begin standing with their toes positioned against a marker. Players initiated the jump with countermovement and arm swing, jumping horizontally as far as possible and landing on both feet. The jump was invalid if the players did not land properly on their feet or fell back.

SECONDARY OUTCOMES:
CMJ | 10 weeks
  Players performed two jumps [19] for each protocol, with one minute of rest provided between trials and three minutes of rest between protocols. The best result was recorded for analysis. CMJ height was calculated with an Optojump system (Microgate, Bolzano, Italy). For the CMJ, participants began by standing upright. Upon readiness, the athlete squatted down until the knees were bent at a 90-degree angle and then immediately executed a vertical jump as high as possible. Throughout the test, participants kept their hands on their hips[20].

OTHER OUTCOMES:
Drop Jump | 10 weeks
  Players performed two jumps [19] for each protocol, with one minute of rest provided between trials and three minutes of rest between protocols. The best result was recorded for analysis. DJ height were calculated with an Optojump system (Microgate, Bolzano, Italy).
  The optimal DJ height was determined in the initial familiarization session. Following preliminary pilot testing, each player performed three DJs from two heights (90 and 110 cm) with 1-min intervals. The highest jump height/contact time ratio was considered the optimal height. In the DJ, the players drop from the optimal with one foot, landing with 2 feet simultaneously, and then immediately perform a maximal jump [21]. The RSI was calculated by dividing flight time (ms) by contact time (ms) [22].
Drop jump (RSI) | 10 weeks
  The RSI was calculated by dividing flight time (ms) by contact time (ms) [22].
Linear sprint-5m | 10 weeks
  Participants performed two 20-m sprints (with 5-m split time also recorded), with at least three minutes of rest between them. The fastest performance trial was used for data analysis. During the recovery period between sprints, the participants returned to the starting line and waited for the second trial. Sprint times were recorded with electronic photocells (Timing-Radio Controlled; TTSport, San Marino, CA, USA) placed 5-m- and 20-m from the starting line. Players were instructed to start the sprints from a line set 0.3-m behind the start line and to run as quickly as possible through the final pair of sensors [19]. During each trial, players were also verbally encouraged to produce their maximal effort.
Linear sprint-20m | 10 weeks
  Participants performed two 20-m sprints (with 5-m split time also recorded), with at least three minutes of rest between them. The fastest performance trial was used for data analysis. During the recovery period between sprints, the participants returned to the starting line and waited for the second trial. Sprint times were recorded with electronic photocells (Timing-Radio Controlled; TTSport, San Marino, CA, USA) placed 5-m- and 20-m from the starting line. Players were instructed to start the sprints from a line set 0.3-m behind the start line and to run as quickly as possible through the final pair of sensors [19]. During each trial, players were also verbally encouraged to produce their maximal effort.
Change of direction | 10 weeks
  The players performed the CODS [23] test to measure the change of direction ability. The players performed two trials separated by three minutes of rest. The fastest of the two trials was used for analysis. Single-beam measure were taken using electronic photocells (Timing-Radio Controlled; TTSport, San Marino, CA, USA) which is previously validated system [24], positioned 3 meters apart and located on either side of the start and finish lines. All photocells were mounted at a height of 1 m above the floor, the maximum height of the manufacturer's standard tripods. The players started the trials from a line placed 0.3-m behind the start line. During each trial, players were strongly verbally encouraged to produce their maximal effort.

CONTACTS AND LOCATIONS:
Locations (1):
- Vytutas Magnus University, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP